CLINICAL TRIAL: NCT03541980
Title: Does IV Acetaminophen Reduce Opioid Requirement in Pediatric Emergency Department Patients With Acute Sickle Cell Crises?
Brief Title: Does IV Acetaminophen Reduce Opioid Requirement in Pediatric Patients With Acute Sickle Cell Crises?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Newark Beth Israel Medical Center (Other)
Responsible Party: Principal Investigator, Cena Tejani, Principal Investigator, Newark Beth Israel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017.48
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Sickle Cell Anemia Crisis
Keywords: sickle cell; acetaminophen in pain crises; opioid-sparing
MeSH Terms: conditions — Vaso-Occlusive Crises | interventions — Acetaminophen; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Active Comparator): Patients allocated to receive IV acetaminophen
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Patients allocated to receive IV normal saline placebo
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Acetaminophen — Administration of 15 mg/kg (1000 mg max dose) of IV acetaminophen
  Other Names: Ofirmev; Tylenol
  Arms: Intervention
Drug: Normal saline — Normal saline volume equivalent
  Other Names: Sodium chloride solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether IV acetaminophen can decrease the need for subsequent opioid administration in the acute management of sickle cell crisis pain in the pediatric emergency room.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, double-blinded, controlled study in an academic urban pediatric emergency department of children with sickle cell disease presenting with acute sickle cell crisis pain between ages of 4 to 16 years, with a pain score of 6/10 or higher on the Wong-Baker modified FACES pain scale. In order to detect a difference of 0.2 mg/kg in cumulative dosage of morphine (at our institution, 0.3 mg/kg morphine deems an inpatient admission for parenteral pain management) with 80% power and alpha of 0.05, we calculated a sample size of 33 patients in each group. All patients will receive IV ketorolac and IV morphine. Patients will be randomized to receive IV acetaminophen or IV saline (volume-equivalent). Pain scores will be obtained at baseline, and again at 30 minutes, 60 minutes, 90 minutes, and 120 minutes after medication administration. Cumulative morphine dosing, rates of admission, and rates of adverse effects of morphine will also be analyzed. Our primary objective is to decrease the need for subsequent opioid administration. Our secondary objectives are to determine if IV Acetaminophen decreases pain score at 30 minutes, 60 minutes, 90 minutes, and 120 minutes, decreases the rate of admissions, and decreases the rate of adverse effects from opioids.

ELIGIBILITY:
Inclusion Criteria:

* Any patient age 4-16 years with sickle cell disease who presents the Pediatric ER with acute sickle cell pain crisis with a pain of 6/10 or higher

Exclusion Criteria:

* Patient with fever (38C or 100.4F)
* Patient less than age 4 years
* Patient greater than age 16 years
* Patient with hypersensitivity/allergy to either morphine, NSAIDs, or acetaminophen
* Patient received acetaminophen within the past 4 hours
* Patient with known liver disease or renal disease
* Patient not requiring IV morphine (pain score 5/10 or less)
* Patient enrolled in the study within the past 72 hours

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cena Tejani, MD, Principal Investigator — Children's Hospital of NJ at Newark Beth Israel Medical Center
Locations (1):
- Newark Beth Israel, Newark, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhebaria T, Sivitz A, Tejani C. Does Intravenous Acetaminophen Reduce Opioid Requirement in Pediatric Emergency Department Patients With Acute Sickle Cell Crises? Acad Emerg Med. 2021 Jun;28(6):639-646. doi: 10.1111/acem.14149. Epub 2020 Oct 30. PMID 33025690

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients allocated to receive IV acetaminophen-35
  Acetaminophen: Administration of 15 mg/kg (1000 mg max dose) of IV acetaminophen
- Placebo: Patients allocated to receive IV normal saline placebo-36
  Normal saline: Normal saline volume equivalent
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 35 | 36
Completed | 35 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 36 | 71
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 21 | 16 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 34 | 68
  White | 0 | 0 | 0
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 36 | 71

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Opioid Dosing
Description: Total dosing of opioid given after initial evaluation in mg/kg
Time Frame: 120 minutes
Measure: Mean (99% Confidence Interval); unit: mg/kg
Groups:
- Intervention: Patients allocated to receive IV acetaminophen
  Acetaminophen: Administration of 15 mg/kg (1000 mg max dose) of IV acetaminophen
  .2mg/kg
- Placebo: Patients allocated to receive IV normal saline placebo
  Normal saline: Normal saline volume equivalent
  .2mg/kg
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 35 | 36
mg/kg | .2 [.1 to .2] | .2 [.1 to .2]

2. Secondary Outcome: Pain Scores
Description: Scale of 1-10 Pain scale, Min value 1, Max value 10, higher score is worse
Time Frame: at disposition
Measure: Mean (99% Confidence Interval); unit: pain intensity measured on scale 1-10
Groups:
- Intervention: Patients allocated to receive IV acetaminophen
  Acetaminophen: Administration of 15 mg/kg (1000 mg max dose) of IV acetaminophen 5.5
- Placebo: Patients allocated to receive IV normal saline placebo
  Normal saline: Normal saline volume equivalent 5.2
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 35 | 36
pain intensity measured on scale 1-10 | 5.5 [4.3 to 6.6] | 5.2 [4.2 to 6.3]

3. Secondary Outcome: Inpatient Admission
Description: Percentage of patients admitted to the inpatient unit for parenteral pain management
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 35 | 36
Participants | 25 | 21

4. Secondary Outcome: Adverse Effects
Description: Rate of adverse effects experienced by patients from opioid administration vs acetaminophen administration
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 35 | 36
Participants | 0 | 0

5. Secondary Outcome: Percentage of the Patients Reporting Satisfaction
Description: How satisfied were patients with the management of their pain
Time Frame: 120 minutes
Measure: Mean (99% Confidence Interval); unit: percent
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 35 | 36
percent | 84 [77.2 to 91.8] | 85 [76.2 to 93.4]

ADVERSE EVENTS:
Time Frame: 120 minutes
Groups:
- Intervention: Patients allocated to receive IV acetaminophen
  Acetaminophen: Administration of 15 mg/kg (1000 mg max dose) of IV acetaminophen
  none
- Placebo: Patients allocated to receive IV normal saline placebo
  Normal saline: Normal saline volume equivalent
  none
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03541980/Prot_SAP_000.pdf